CLINICAL TRIAL: NCT04544943
Title: A Randomised, Double-Blind, Vehicle Controlled, Sequential Group Study to Determine the Safety, Tolerability, Pharmacokinetics and Efficacy of Twice Daily Application of Topical BioLexa in Adult Healthy Subjects and Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of Twice Daily Application of Topical BioLexa in Adult Healthy Subjects and Patients With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoth Therapeutics, Inc. (Other)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-001
Record Dates: First submitted 2020-08-27; First posted 2020-09-10 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Route of Administration: Topical; Dosage Form: Topical lotion. Product Name: BioLexa. The total body surface area (BSA) dosed will be either 9% or 27% BSA. Part A will include both an active-control (lotion base + 0.1% gentamicin) and a placebo control, applied at 9% or 27% BSA.
  Interventions: Drug: BioLexa- Cohort 1; Drug: Placebo; Drug: Gentamicin
- Cohort 2 (Placebo Comparator): Route of Administration: Topical; Dosage Form: Topical lotion. Product Name: BioLexa. The minimum % BSA dosed will be 3% BSA and the maximum will be 27% BSA for patients in Cohort 2. Part B will include both an active-control (lotion base + 0.1% gentamicin) and a placebo control.
  Interventions: Drug: BioLexa- Cohort 2; Drug: Placebo; Drug: Gentamicin
- Open-Label (Experimental): Route of Administration: Topical; Dosage Form: Topical lotion. Product Name: BioLexa. The minimum % BSA dosed will be 3% BSA and the maximum will be 27% BSA for patients
  Interventions: Drug: BioLexa- Cohort 1

INTERVENTIONS:
Drug: BioLexa- Cohort 1 — Twice daily application of topical BioLexa™ lotion, administered for 14 days in adult healthy subjects
  Arms: Cohort 1; Open-Label
Drug: BioLexa- Cohort 2 — Twice daily application of topical BioLexa™ lotion, administered for 14 days in adult mild to moderate AD patients
  Arms: Cohort 2
Drug: Placebo — Twice daily (BID) application of placebo for 14 days
  Arms: Cohort 1; Cohort 2
Drug: Gentamicin — Twice daily (BID) application of Gentamicin for 14 days
  Arms: Cohort 1; Cohort 2

SUMMARY:
This is a Phase 1, randomised, double-blind, vehicle controlled study to determine the safety, tolerability, PK and efficacy of twice daily application of topical BioLexa™ lotion, administered for 28 days in adult healthy subjects, in adult patients with mild to moderate AD and in adolescent patients with mild to moderate AD.

DETAILED DESCRIPTION:
This study will consist of 3 parts. Part A: Part A will consist of Cohort 1 constituting of heathy subjects. The total body surface area (BSA) dosed will be either 9% or 27% BSA for Cohort 1 subjects. Part A will include both an active-control (lotion base + 0.1% gentamicin) and a placebo control, applied at 9% or 27% BSA.

Part B: Part B will consist of Cohort 2 made up of adult mild to moderate AD patients. The minimum %BSA dosed will be 3% BSA and the maximum will be 27% BSA for patients in Cohort 2. Part B will include both an active-control (lotion base + 0.1% gentamicin) and a placebo control.

Open-Label Cohort: After closure of Part B, open-label enrolment of patients with mild to moderate atopic dermatitis affecting 3-27% BSA for treatment with BioLexa for 14 days (unblinded).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers, aged 18 to 65 years
2. Participants must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of study drug; (Part A)
3. Participants must have a BMI between ≥ 18.0 and ≤ 35.0 kg/m2 at Screening; (Part A and B)
4. Participants must have clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or delegate; (Part A and B)
5. Participants must be a non-smoker or a smoker who smokes no more than 2 cigarettes or equivalent per week in order to be included in the study; (Part A and B)
6. Participants must have no relevant dietary restrictions, and be willing to consume standard meals provided; (Part A and B)
7. Females must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from screening until study completion, including the follow-up period.
8. Males must not donate sperm for at least 90 days after the last dose of study drug (Part A and B);
9. Participants must have the ability and willingness to attend the necessary visits to the CRU (Part A and B);
10. Participants must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures (Part A and B).

    In addition to the above-mentioned criteria, participants in Part B should also fulfill the following inclusion criteria:
11. Male and Female, 18 to 65 years (Cohort 2 - adult patients)
12. Physician documented history or confirmed diagnosis of mild to moderate AD for at least 6 months prior to screening. AD should be diagnosed by EASI score of Mild or Moderate on Day 1;
13. Mild to moderate AD with a minimum of 3% to a maximum of 27% BSA involvement on Day 1 (excluding the scalp, designated venous access areas, palms and soles);
14. Participant has a minimum of 2 AD lesions;
15. Informed consent of parent(s) or legal guardian, and, if age appropriate, assent by the patient, as required by local laws;

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period; (Part A and B)
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant; (Part A and B)
3. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol; (Part A and B)
4. Blood donation or significant blood loss within 60 days prior to the first study drug administration; (Part A and B)
5. Plasma donation within 7 days prior to the first study drug administration; (Part A and B)
6. Fever (body temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening; (Part A and B)
7. History of severe allergic or anaphylactic reactions; (Part A and B)
8. Known contact sensitivity to aminoglycosides; (Part A and B)
9. Contact sensitivity to BioLexa or any formulation ingredients; (Part A and B)
10. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening; (Part A and B)
11. Abnormal ECG findings at Screening that are considered by the Investigator to be clinically significant; (Part A and B)
12. History or presence of a condition associated with significant immunosuppression; (Part A and B)
13. History of life-threatening infection (e.g. meningitis); (Part A and B)
14. Infections requiring parenteral antibiotics within the 6 months prior to Screening; (Part A and B)

    In addition to the above-mentioned criteria, participants in Part B who also fulfill the following exclusion criteria must be excluded from the study:
15. Have used antiseptic treatments (e.g. bleach baths, potassium permanganate etc.) within 1 month before Baseline visit. (Patients who have recently used antiseptic treatment may be rescreened at a later date if they wish to participate in the study and agree to stop antiseptic treatment)
16. Treatment with the following topical agents within 2 weeks before the Baseline visit: corticosteroids, phosphodiesterase inhibitors, tacrolimus or pimecrolimus.
17. Systemic treatment for AD or for condition, with steroids or other immunosuppressive/immunomodulating substances, e.g., cyclosporine, mycophenolate-mofetil, azathioprine or methotrexate within 4 weeks before the Baseline visit or 5 half-lives whichever is longer. Use of steroid inhalers and nasal corticosteroids is allowed
18. Treatment with any cell depleting agents, e.g., rituximab, within 6 months of the Baseline visit or treatment with other biologics within 3 months of the Baseline visit
19. Prior treatment with dupilumab or any antibody against IL-4Rα or IL-13 within 1 month before Baseline visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) of BioLexa™ and active control (gentamicin only) | Measurements at Baseline till Follow-up/EOS visit (14 days) or early termination
  Measured by Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of BioLexa™ and active control (gentamicin only) in patients with mild to moderate AD (Part B only)- by Eczema Area and Severity Index (EASI) score | Measured on Day 7, 14, 21 and 28
  Measured by the change from Baseline in the Eczema Area and Severity Index (EASI) score
To evaluate the preliminary efficacy of BioLexa™ in patients with mild to moderate AD (Part B only)- by Scoring Atopic Dermatitis | Measured on on Day 7, 14, 21 and 28
  Measured by the change from Baseline in Scoring Atopic Dermatitis (SCORAD) index
To characterize pharmacokinetic (PK) profile of BioLexa and active control (gentamicin only) (Part A and B)- AUC | Measurements at Baseline till the end of the study (14 days)
  Measured through Area under the curve (AUC)
To characterize pharmacokinetic (PK) profile of BioLexa and active control (gentamicin only) (Part A and B)- Cmax | Measurements at Baseline till the end of the study (14 days)
  Measured through maximum (or peak) serum concentration (Cmax)
To characterize pharmacokinetic (PK) profile of BioLexa and active control (gentamicin only) (Part A and B)- Tmax | Measurements at Baseline till the end of the study (14 days)
  Measured through time of peak concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cumming, Dr, Principal Investigator — Novatrials
Locations (1):
- Novatrials, Kotara, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No